CLINICAL TRIAL: NCT07108465
Title: Comparative Experimental Study Between Bupivacaine and Ropivacaine Regarding Efficacy in Third Molar Removal Surgery Under General Anesthesia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Henrique Tedesco (Other)
Responsible Party: Sponsor-Investigator, Henrique Tedesco, Principal Investigator, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 89726325.2.0000.5327
Record Dates: First submitted 2025-07-22; First posted 2025-08-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-08

CONDITIONS: Third Molars Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Bupivacaine (Active Comparator): use of bupivacaine 0,5% + epinephrine 0,2mL in third molar surgery in general anesthesia
  Interventions: Drug: Bupivacaine 0,5%
- Group B - Ropivacaine (Active Comparator): use of ropivacaine 0,75% + epinephrine 0,2mL in third molar surgery in general anesthesia
  Interventions: Drug: Ropivacaine 0,75%

INTERVENTIONS:
Drug: Bupivacaine 0,5% — Injection of bupivacaine 0,5% in group A
  Arms: Group A - Bupivacaine
Drug: Ropivacaine 0,75% — Injection of ropivacaine 0,75% in group B
  Arms: Group B - Ropivacaine

SUMMARY:
The goal of this clinical trial is to compare the efficacy of bupivacaine and ropivacaine in third molar removal surgery under general anesthesia in healthy volunteers. The main question aims to determine whether there is any difference in vital signs, hemostasis and postoperative pain between ropivacaine and bupivacaine in patients undergoing third molars extraction under general anesthesia.

Researchers will compare bupivacaine and ropivacaine in a split-mouth study to determine if one drug is more effective in third molar extraction surgery under general anesthesia (better hemostasis, less postoperative pain, and fewer changes in vital signs). Participants will undergo a single surgical procedure and complete the Visual Analog Scale to record postoperative pain

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 60
* Patients ASA Physical Status Classification I and II
* Patients with impacted or semi-impacted lower third molars with similar positioning on both sides according to the Pell and Gregory classification

Exclusion Criteria:

* Patients who can have surgery under local anesthesia
* Patients where more procedures are required in the same surgical session

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate if there is a significant difference between groups in postoperative analgesic capacity using Visual Analog Scale, intraoperative hemostasis and in vital signs during anesthesia. | From surgery to 7 postoperative days
  The Visual Analog Scale (0-10 VAS) can be interpreted as no pain (0), mild (1-3), moderate (4-6),severe (7-9),or worse pain (10)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalath RN, Kulal R, Gopinath S. Comparison of clinical efficacy of ropivacaine and lignocaine with adrenaline for implant surgery anesthesia: a split-mouth randomized controlled clinical trial. J Dent Anesth Pain Med. 2021 Aug;21(4):337-344. doi: 10.17245/jdapm.2021.21.4.337. Epub 2021 Jul 30. PMID 34395901

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT07108465/Prot_ICF_000.pdf